CLINICAL TRIAL: NCT07062757
Title: The Effect of Lymphatic Drainage Massage and Melatonin on Pain and Edema After Orthognathic Surgery.
Brief Title: Lymphatic Drainage Massage and Melatonin in Post-Orthognathic Surgery Pain and Edema
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-190312
Record Dates: First submitted 2025-06-30; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dentofacial Deformities; Edema; Pain
Keywords: dentafacial deformities; edema; pain
MeSH Terms: conditions — Dentofacial Deformities; Edema; Pain | interventions — Manual Lymphatic Drainage; Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (No intervention) (Sham Comparator): No intervention will be applied to prevent edema in this group of patients.
  Interventions: Other: no intervention
- group 2 (lymphatic drainage massage) (Experimental): In this group of patients, a total of 10 sessions of lymphatic drainage massage will be applied, starting from the 2nd postoperative day, with 2 sessions per week
  Interventions: Other: lymphatic drainage massage
- group 3 (oral melatonin tablet) (Experimental): In this group of patients, the first dose of 10 mg oral melatonin tablet will be administered one day before the operation, and the patients will take the tablet daily for a total of 21 days.
  Interventions: Dietary Supplement: oral melatonin tablet
- group 4 (both melatonin and lymphatic drainage) (Experimental): In this group of patients, both melatonin and lymphatic drainage procedures will be applied together.
  Interventions: Other: lymphatic drainage massage; Dietary Supplement: oral melatonin tablet; Combination Product: both melatonin and lymphatic drainage

INTERVENTIONS:
Other: no intervention — this group patients receive any medication for edema control.
  Arms: group 1 (No intervention)
Other: lymphatic drainage massage — A total of 10 sessions of lymphatic drainage massage will be applied to this group of patients, starting from the 2nd postoperative day, with 2 sessions per week.
  Arms: group 2 (lymphatic drainage massage); group 4 (both melatonin and lymphatic drainage)
Dietary Supplement: oral melatonin tablet — In this group of patients, the first dose of 10 mg oral melatonin tablet will be given one day prior to the operation, and the patients will continue taking the tablet daily for a total of 21 days.
  Arms: group 3 (oral melatonin tablet); group 4 (both melatonin and lymphatic drainage)
Combination Product: both melatonin and lymphatic drainage — In this group of patients, a total of 10 sessions of lymphatic drainage massage will be applied starting from the 2nd postoperative day, with 2 sessions per week, while the first dose of 10 mg oral melatonin tablet will be administered one day prior to the operation, and the patients will continue taking the tablet daily for 21 days.
  Arms: group 4 (both melatonin and lymphatic drainage)

SUMMARY:
Lymphatic drainage massage is one of the most essential techniques for reducing edema. It is a very gentle, monotonous, slow, rhythmic massage applied to the skin's surface. This technique accelerates the flow of lymphatic fluid, minimizing swelling and providing relief. Frequently used after orthognathic surgery, lymphatic drainage massage helps reduce edema, enhancing patients' postoperative comfort.

DETAILED DESCRIPTION:
Melatonin, a hormone produced by the pineal gland, is a neurochemical substance that functions in harmony with the body's natural rhythm. In addition to its presence in the brain, melatonin can also be found in the retina, bone marrow, intestines, skin, and various blood cells. Conditions such as insomnia or jet lag may benefit from melatonin supplements. Beyond its role in improving sleep quality, melatonin also contributes to regulating the immune system, body temperature, blood pressure, and cortisol hormone levels.

Another important function of melatonin is its powerful free radical-scavenging ability. It can neutralize both reactive oxygen species and reactive nitrogen species. Due to its strong antioxidant properties, several studies have investigated its effects on pain and edema. Research has shown that preoperative and postoperative melatonin administration can reduce postoperative pain and accelerate sensory recovery through its antioxidant effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dentofacial deformities who are planned to undergo orthognathic surgery
2. Patients who have not previously undergone orthognathic surgery
3. Patients with no systemic diseases

Exclusion Criteria:

1. Presence of systemic diseases affecting general health
2. Presence of malignant disease in the head and neck region
3. Patients who have previously undergone orthognathic surgery
4. Patients with any bleeding disorders
5. Patients with cardiovascular disease who are under anticoagulant or antiplatelet therapy

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative edema assessment | 1month
  Postoperative edema measurements will be taken after the patient is anesthetized before surgery and on the 1st, 3rd, and 7th postoperative days. Before the surgery, the gonion and tragus will be marked with methylene blue, and the distance between the gonion-lateral canthus and tragus-labial commissure will be measured and recorded using a thread. Measurements will be repeated on postoperative days 1, 3, 7, 14, 21, and 28 and recorded in the evaluation form.

SECONDARY OUTCOMES:
pain assessment | 1 month
  VAS assessment will be performed on all days when edema measurements are taken for pain evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)